CLINICAL TRIAL: NCT03436329
Title: Reduced Dissemination of Tumor Cells With Primary Ligation of the Vein in Patients With Lung Cancer: A Multi-centre Randomized Controlled Trial
Brief Title: Reduced Dissemination of Tumor Cells With Primary Ligation of the Vein in Patients With Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Lunxu Liu, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TSCI005
Record Dates: First submitted 2018-02-05; First posted 2018-02-19 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Lung Cancer; Surgery; Circulating Tumor Cell
Keywords: Lung cancer; Surgical technique; vessel ligation; Circulating tumor cell
MeSH Terms: conditions — Lung Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vein ligation first (Experimental): During this procedure, patients undergo lobectomy with the pulmonary vein ligated first.
  Interventions: Procedure: Vein ligation first
- Artery ligation first (Active Comparator): During this procedure, patients undergo lobectomy with the pulmonary artery ligated first.
  Interventions: Procedure: Artery ligation first

INTERVENTIONS:
Procedure: Vein ligation first — During this procedure, patients undergo lobectomy with the pulmonary vein ligated first.
  Arms: Vein ligation first
Procedure: Artery ligation first — During this procedure, patients undergo lobectomy with the pulmonary artery ligated first.
  Arms: Artery ligation first

SUMMARY:
The purpose of this study is to assess the impact of the sequence of vessel interruption in lung cancer patients on tumor cell spread and patient survival by using peripheral blood circulating tumor cells.

DETAILED DESCRIPTION:
Circulating tumor cells (CTCs) in the peripheral blood can be a biomarker to predict tumor recurrence and survival. Handling the tumor during a surgery may promote the release of CTCs into the bloodstream. Therefore, in a surgery of cancer, interruption of the vein before ligation of the artery may be justified. This multi-center randomized controlled trial is to assess the impact of the sequence of vessel interruption in lung cancer patients on tumor cell spread and patient survival by using peripheral blood CTCs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage I-IV lung cancer eligible for surgery
2. Patients undergoing the completely thoracoscopic lobectomy
3. The nodule size was more than 2.5 cm
4. Patients consenting for intraoperative blood sampling

Exclusion Criteria:

1. Patients who underwent primary wedge resection and open lobectomy
2. Patients who received neoadjuvant therapy before surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The changes of the level of circulating tumor cells in the peripheral blood | Intraoperative
  The changes of the level of circulating tumor cells in the peripheral blood before cutting the skin and after closing the chest

SECONDARY OUTCOMES:
3-year Progression-Free-Survival | From date of the recruitment, assessed up to 36 months
  From the date of recruitment until the date of progression of lung cancer assessed up to 36 months
Blood loss | During the surgery
  Blood loss during the surgery
Operative time | During the surgery
  Operative time during the surgery
Length of stay | From date of admission until the date of discharging or date of death from any cause in hospital, whichever came first, assessed up to 30 days
  The length of patients staying in hospital from the date of checking in to the date of checking out
Morbidity | Within 30 days after surgery
  Complications resulting from surgery, such as pneumonia, air leak and arrhythmia.

CONTACTS AND LOCATIONS:
Overall Officials: Lunxu Liu, M.D.,Ph.D., Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gall TM, Jacob J, Frampton AE, Krell J, Kyriakides C, Castellano L, Stebbing J, Jiao LR. Reduced dissemination of circulating tumor cells with no-touch isolation surgical technique in patients with pancreatic cancer. JAMA Surg. 2014 May;149(5):482-5. doi: 10.1001/jamasurg.2013.3643. PMID 24599353
- [Background] Hansen E, Wolff N, Knuechel R, Ruschoff J, Hofstaedter F, Taeger K. Tumor cells in blood shed from the surgical field. Arch Surg. 1995 Apr;130(4):387-93. doi: 10.1001/archsurg.1995.01430040049007. PMID 7710337
- [Background] Li F, Jiang G, Chen Y, Wang J. Curative Effects of Different Sequences of Vessel Interruption During the Completely Thoracoscopic Lobectomy on Early Stage Non-Small Cell Lung Cancer. Ann Thorac Cardiovasc Surg. 2015;21(6):536-43. doi: 10.5761/atcs.oa.15-00044. Epub 2015 Aug 18. PMID 26289504
- [Background] Kozak A, Alchimowicz J, Safranow K, Wojcik J, Kochanowski L, Kubisa B, Pierog J, Grodzki T. The impact of the sequence of pulmonary vessel ligation during anatomic resection for lung cancer on long-term survival--a prospective randomized trial. Adv Med Sci. 2013;58(1):156-63. doi: 10.2478/v10039-012-0061-3. PMID 23612700
- [Background] Refaely Y, Sadetzki S, Chetrit A, Simansky DA, Paley M, Modan B, Yellin A. The sequence of vessel interruption during lobectomy for non-small cell lung cancer: is it indeed important? J Thorac Cardiovasc Surg. 2003 Jun;125(6):1313-20. doi: 10.1016/s0022-5223(03)00022-9. PMID 12830050
- [Background] Kurusu Y, Yamashita J, Hayashi N, Mita S, Fujino N, Ogawa M. The sequence of vessel ligation affects tumor release into the circulation. J Thorac Cardiovasc Surg. 1998 Jul;116(1):107-13. doi: 10.1016/s0022-5223(98)70248-x. PMID 9671904
- [Background] Ge MJ, Shi D, Wu QC, Wang M, Li LB. Observation of circulating tumour cells in patients with non-small cell lung cancer by real-time fluorescent quantitative reverse transcriptase-polymerase chain reaction in peroperative period. J Cancer Res Clin Oncol. 2006 Apr;132(4):248-56. doi: 10.1007/s00432-005-0059-3. Epub 2005 Dec 1. PMID 16320073
- [Background] Yellin A, Sadetzki S, Simansky DA, Refaely Y, Chetrit A, Paley M. The sequence of vessel interruption during lobectomy: does it affect the amount of blood retained in the lobe? Eur J Cardiothorac Surg. 2007 Apr;31(4):711-3. doi: 10.1016/j.ejcts.2007.01.019. Epub 2007 Feb 15. PMID 17306554
- [Background] Hashimoto M, Tanaka F, Yoneda K, Takuwa T, Matsumoto S, Okumura Y, Kondo N, Tsubota N, Tsujimura T, Tabata C, Nakano T, Hasegawa S. Significant increase in circulating tumour cells in pulmonary venous blood during surgical manipulation in patients with primary lung cancer. Interact Cardiovasc Thorac Surg. 2014 Jun;18(6):775-83. doi: 10.1093/icvts/ivu048. Epub 2014 Mar 11. PMID 24618055
- [Background] Song PP, Zhang W, Zhang B, Liu Q, DU J. Effects of different sequences of pulmonary artery and vein ligations during pulmonary lobectomy on blood micrometastasis of non-small cell lung cancer. Oncol Lett. 2013 Feb;5(2):463-468. doi: 10.3892/ol.2012.1022. Epub 2012 Nov 9. PMID 23420582
- [Background] Ackerman NB. Primary arterial ligation in resection of cancer of the colon. Rational and technic. Am J Surg. 1977 Jan;133(1):73-7. doi: 10.1016/0002-9610(77)90196-9. PMID 835783
- [Derived] Wei S, Guo C, He J, Tan Q, Mei J, Yang Z, Liu C, Pu Q, Ma L, Yuan Y, Lin F, Zhu Y, Liao H, Wang W, Liu Z, Li Q, Jiang B, Li C, Xia L, Zhao K, Gan F, Cheng J, Wu Z, Wang Y, Lin Y, Kou Y, Che G, Chen L, Li J, Liu L. Effect of Vein-First vs Artery-First Surgical Technique on Circulating Tumor Cells and Survival in Patients With Non-Small Cell Lung Cancer: A Randomized Clinical Trial and Registry-Based Propensity Score Matching Analysis. JAMA Surg. 2019 Jul 1;154(7):e190972. doi: 10.1001/jamasurg.2019.0972. Epub 2019 Jul 17. PMID 31042283